CLINICAL TRIAL: NCT06324487
Title: Blood Flow Restrictive Exercise Application in the Treatment of Subacromial Impingement Syndrome
Brief Title: A New Application in Subacromial Impingement Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Nursena Cansabuncu, MSc candidate, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-772.02-7487
Record Dates: First submitted 2024-02-26; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Subacromial Impingement Syndrome
Keywords: subacromial impingement syndrome; rehabilitation; exercise
MeSH Terms: conditions — Shoulder Impingement Syndrome; Motor Activity | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SEP Group (Active Comparator): The treatment will be individualized by calculating the appropriate resistance loads for the exercise program. All participants will undergo progressive exercises in sessions conducted by a physiotherapist.
  Interventions: Other: Progressive Exercises
- BFRT Group (Experimental): People in the BFRT categories will perform the exercise program at approximately 20-30% resistance of 1-RM, and an upper arm reinforcement occlusion cuff will be used during strengthening exercises with dumbbells for the rotator cuff and scapula girdles
  Interventions: Other: Progressive Exercises; Other: Blood Flow Restriction Therapy

INTERVENTIONS:
Other: Progressive Exercises — Electrotherapy, stretching of the capsules, strengthening, ROM exercises, proprioceptive exercises
Other: Blood Flow Restriction Therapy — Strengthening exercises performed by using cuff surrounding proximal part of the arm.
  Arms: BFRT Group

SUMMARY:
Individuals diagnosed with Subacromial Impingement Syndrome by a physical therapist based on MRI results and examination findings will be included in the study. 40 people will be randomly divided into blood flow restrictive exercise (BFRT) and structured exercise program (SEP) groups, 20 people in each group. Participants will receive two evaluations: before starting treatment and immediately after 4 weeks of treatment. Pain, shoulder ROM, shoulder functional level, quality of life, shoulder muscle strength, grip strength, and sleep quality evaluation will be performed. The treatment program will be 5 days a week for a total of 4 weeks. The treatment will be individualized by calculating the appropriate resistance loads for the exercise program. All participants will undergo progressive exercises in sessions conducted by a physiotherapist.

DETAILED DESCRIPTION:
The study is planned to be carried out between September 2023 and June 2024. Individuals diagnosed with Subacromial Impingement Syndrome by a physical therapist based on MRI results and examination findings will be included in the study. The sample size of this study was calculated using G-Power 3.1.9.7. Assuming that effect sizes (ES) are 0.99, significance level (a) is 0.05, and statistical power (1-b) is 0.8, a minimum of 36 participants in total are required for this study. Considering the 10% dropout rate, it is planned to include 40 people in our study. The 40 people included will be randomly divided into blood flow restrictive exercise (BFRT) and structured exercise program (SEP) groups, with 20 people in each group. Randomization will be generated using the random number sequence www.random.org.

Criteria for Inclusion in the Study

* Being Volunteer
* Being between the ages of 25-65
* Being diagnosed with Stage 2 or 3 Subacromial Impingement Syndrome
* Not having had a steroid injection in the last 6 months

Exclusion Criteria from the Study

* Having neuromuscular disease
* History of upper extremity fracture
* Cardiovascular diseases
* Rheumatic diseases
* Having had shoulder, neck, elbow or hand surgery
* Presence of acute inflammation

Evaluation Methods Demographic Information Form: In order to collect demographic information, a form that questions age, gender, height, weight, occupation, education level, smoking, alcohol and substance use, city of residence and previous counseling or alternative treatment history has been created and is presented in the appendix.Participants will receive two evaluations: before starting treatment and immediately after 4 weeks of treatment.

Pain assessment: It will be made with Visual Analog Scale (VAS). VAS is a scale that provides patient-based measurement between the perception of "painless" and "most severe pain" in a vertical or horizontal plane with a length of 10 cm divided into equal intervals. Individuals will be asked to mark on the scale the degree of pain they feel at rest, during arm elevation and during sleep, on a 10 cm line.

Shoulder ROM Evaluation: It will be done with a universal goniometer. Individuals' shoulder flexion, abduction, internal and external range of motion will be evaluated actively and passively while in the supine position.

Shoulder Functional Level Evaluation: It will be done with the Quick Disability Scale of the Arm, Shoulder and Hand (Quick-DASH). The Arm, Shoulder and Hand Disability Scale (DASH) is a tool developed to assess the health status of patients with upper extremity disorders. Shorter surveys are preferred because they are easy to understand and can be completed quickly by patients. In this context, DASH is abbreviated as Quick DASH, the 11-item Quick Disability of the Arm, Shoulder and Hand questionnaire. It was developed to measure physical function and symptoms in patients with upper extremity disorders. The survey consists of 11 items. Answers are scored from 1 (no difficulty) to 5 (not able to do it at all). A total score of 100 was expressed as the highest disability, while a total score of 0 indicated no disability. Turkish validity and reliability were evaluated by Evcik et al. It was made by in 2011.

Quality of Life Assessment: It will be done with the short form (SF-36). SF-36 is a test consisting of 36 items that the person fills out and answers himself to obtain information about the person's health status. It consists of 8 sub-parameters: physical function, physical role difficulty, emotional role difficulty, pain, mental health, social functionality, energy/vitality/vitality, and general health perception. Turkish validity and reliability were determined by Koçyiğit et al. It was made by in 1999.

Shoulder Muscle Strength Assessment: A hand dynamometer will be used to evaluate the shoulder flexor, abductor, internal rotator and external rotator muscles. The patient and the muscle to be tested will be adjusted to the correct testing position. The dynamometer will be placed distal to the joint at a comfortable level and the patient will actively participate in the evaluation.

Grip Strength Evaluation: The maximum isometric contraction strength of the hand and forearm muscles will be tested. Grip strength is evaluated with the patient in a sitting position. Elbows are kept close to the body and 90 degrees flexed. The patient is asked to grasp the dynamometer and squeeze it as hard as he can. The result of the test is determined by calculating the average of three measurements.

Sleep Quality Assessment: Sleep quality will be evaluated with the Pittsburgh Sleep Quality Index (PSQI). PSQI is a self-report scale consisting of 19 items that evaluates sleep quality and disturbance over the past month. It consists of 24 questions, 19 questions are self-report questions, 5 questions are answered by the spouse or roommate. The 18 scored questions of the scale consist of 7 components (Subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills and daytime dysfunction). Each component is evaluated on a scale of 0-3 points. The total score of the 7 components gives the scale total score. Total score varies between 0-21. A total score greater than 5 indicates "poor sleep quality". Turkish validity and reliability were determined by Ağargün et al. It was made by in 1996.

Treatment Program The treatment program will be planned under the supervision of a physiotherapist, 5 days a week for a total of 4 weeks. The treatment will be individualized by calculating the appropriate resistance loads for the exercise program. All participants will undergo progressive exercises in sessions conducted by a physiotherapist.

In the sessions, before exercise, both groups were given: 80 Hz to the shoulder area for 20 minutes. Electrotherapy will be applied as Asymmetric Biphasic TENS + Hotpack and 1.0 watt/cm2 Ultrasound (US) for 7 minutes.

Exercises to be Performed in Week 1 Shoulder isometric exercises (10 repetitions) Wand exercises for shoulder ROM (Shoulder flexion, abduction, hyperextension, internal and external rotation 10 repetitions) Finger ladder for shoulder ROM (Shoulder flexion and abduction 5 repetitions) Codman exercises for shoulder ROM (10 repetitions) Posterior, anterior and inferior capsule stretches (10 repetitions)

Exercises to be Added in Week 2 Strengthening exercises with dumbbells for the muscles around the rotator cuff and scapula (Shoulder flexion, abduction, external and internal rotation, scapular retraction exercises) (10 repetitions)

Exercises to be Added in Week 3 Pectoral muscle stretching exercise (10 repetitions) Proprioception exercises with a ball on the wall (10 repetitions)

Exercises to be Added in Week 4 Push-up exercise on the wall (10 repetitions) Dynamic stabilization exercise on balance board (10 repetitions)

Strengthening exercises will be applied at different intensities to the BFRT and YEP groups, to which the participants are randomly divided. People in the BFRT group will apply the structured exercise program at approximately 20-30% resistance of 1-RM, and an occlusion cuff surrounding the upper arm will be used during strengthening exercises with dumbbells for the rotator cuff and scapula muscles.

An exercise program consisting of 75 repetitions will be applied throughout four exercise sets, with 30 repetitions in the first set and 15 repetitions in each subsequent set. Rest periods between sets are determined as 30 seconds and the cuff will not be deflated between sets.

Set 1: 30 reps, rest time: 30 seconds Set 2: 15 reps, rest time: 30 seconds Set 3: 15 reps, rest time: 30 seconds Set 4: 15 reps

Determination of Arterial Occlusion Pressure The study will use a personalized tourniquet pressure set at 50% of the limb occlusion pressure according to BFR standards. Patients will be asked to lie on their back while resting comfortably. A vascular Doppler probe (DV-600; Marted, São Paulo, Brazil) will be placed over the brachial artery to capture the auscultatory pulse. To determine the cuff pressure required for complete blood flow restriction, an air cuff will be placed on the patient's arm and then inflated to the point where the auscultatory pulse ceases. This pressure will be recorded as AOP.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 25-65
* Being diagnosed with Stage 2 or 3 Subacromial Impingement Syndrome
* Not having had a steroid injection in the last 6 months

Exclusion Criteria:

* Having neuromuscular disease
* History of upper extremity fracture
* Cardiovascular diseases
* Rheumatic diseases
* Having had shoulder, neck, elbow or hand surgery
* Presence of acute inflammation

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain İntensity | 4 weeks
  The severity shoulder pain was questioned with the Visual Anolog Scale (VAS). The assessment was based on a horizontal 10 cm scale from 1 (least pain) to 10 (the worst pain ever)
Shoulder ROM | 4 weeks
  Shoulder ROM was questioned with the Universal Goniometer. Shoulder flexion, abduction, internal and external range of motion of the individuals in the supine position will be evaluated as active and passive.

SECONDARY OUTCOMES:
Quality of Life Assessment | 4 weeks
  Quality of life assessment was questioned with the Short form-36 (SF-36). SF-36 is a test consisting of 36 items that the person fills out and answers in order to obtain information about the person's health status. It consists of 8 subparameters: international function, physical role strength, emotional role strength, pain, mental health, social functionality, energy/vitality and general health perception.
Sleep Quality Assessment | 4 weeks
  Sleep Quality Assessment was questioned with the Pittsburgh Sleep Quality Index. PSQI is a self-report performance consisting of 19 items that evaluates sleep temperature and disturbance over the past month. It consists of 24 questions, 19 questions are self-report questions, 5 questions are answered by the spouse or roommate. The 18 scored items of the scale are presented with 7 (Subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills and daytime dysfunction). Unites it on 0-3 points. The total score of the 7 components gives the total score. Total score varies between 0-21. A total score greater than 5 indicates "poor sleep standards".
Shoulder Functional Level Assessment | 4 weeks
  Shoulder Functional Level Assessment was questioned with the Quick Disabilities of Arm, Shoulder & Hand. It was developed to measure physical function and symptoms in patients with upper extremity disorders. The survey consists of 11 items. Answers are scored from 1 (no difficulty) to 5 (not able to do it at all). A total score of 100 was expressed as the highest disability, while a total score of 0 indicated no disability.
Shoulder Muscle Strength Assessment | 4 weeks
  A hand dynamometer was used to evaluate the shoulder flexor, abductor, internal rotator and external rotator muscles. The patient and the muscle to be tested will be adjusted to the correct testing position. By adding a dynamometer, the distal part will be placed comfortably and the patient will actively participate in the evaluation.
Grip Strength Assessment | 4 weeks
  Maximum isometric contraction strength of hand and forearm muscles was tested. Grip strength is evaluated with the patient in a sitting position. Elbows are kept close to the body and 90 degrees flexed. The patient is asked to grasp the dynamometer and squeeze it as hard as he can. The result of the test is determined by calculating the average of three measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No